CLINICAL TRIAL: NCT03056599
Title: Feasibility of Assessing Drug Response to Precise Local Injection of Anti-cancer Drugs Using Presage's CIVO Device in Soft Tissue Sarcoma Patients Undergoing Surgery.
Brief Title: Precise Local Injection of Anti-cancer Drugs Using Presage's CIVO Device in Soft Tissue Sarcoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Presage Biosciences (Industry)
Collaborators: Fred Hutchinson Cancer Center (Other); University of Washington (Other); Northwell Health (Other); Oregon Health and Science University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: PRS-2
Record Dates: First submitted 2017-01-22; First posted 2017-02-17 (Actual); Last update posted 2021-09-24 (Actual); Status verified 2021-09

CONDITIONS: Soft Tissue Sarcoma Adult
Keywords: in vivo drug sensitivity; personalized medicine; precision oncology; in vivo oncology; soft tissue sarcoma; chemotherapy; microinjection; microdosing; tumor microenvironment; multiplexed immunohistochemistry
MeSH Terms: conditions — Sarcoma | interventions — Doxorubicin; Docetaxel; Gemcitabine; Interferon-gamma; pembrolizumab; Ipilimumab; Interferon alpha-2; Bortezomib; aldesleukin; Trabectedin; eribulin; olaratumab; atezolizumab; durvalumab; avelumab; Nivolumab; larotrectinib; entrectinib; avapritinib; Sodium Chloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Multiple drug microinjection (Experimental): Patients who are scheduled for surgical biopsy or tumor resection surgery will be injected 4 to 72 hours prior to surgery using the CIVO device. Minute volumes (up to 8.3 microliters) of saline (negative control) or microdoses of anti-cancer agents will be percutaneously injected in a columnar fashion through each of 8 needles into a single enlarged solid tumor.
  Interventions: Drug: Multiple drug microinjection; Device: CIVO device

INTERVENTIONS:
Drug: Multiple drug microinjection — This is a feasibility study in patients with localized or metastatic soft tissue sarcoma undergoing surgery to determine how sarcoma in situ responds to injected microdoses of anti-cancer therapeutics.
  Other Names: Doxorubicin; Docetaxel; Gemcitabine; Interferon gamma; Pembrolizumab; Ipilimumab; Interferon alfa-2B; Bortezomib; Aldesleukin; Trabectedin; Eribulin; Olaratumab; Atezolizumab; Durvalumab; Avelumab; Nivolumab; Larotrectinib; Entrectinib; Avapritinib; Saline
Device: CIVO device — Feasibility of assessing drug response to precise local injection of anti-cancer drugs using Presage's CIVO device in soft tissue sarcoma patients undergoing surgery.

SUMMARY:
This is a feasibility study in patients with localized or metastatic soft tissue sarcoma undergoing surgery to determine how sarcoma in situ responds to injected microdoses of anti-cancer therapeutics.

DETAILED DESCRIPTION:
This is a single arm, pilot study designed to test the feasibility of using the CIVO (Comparative In Vivo Oncology) system in patients with soft tissue sarcoma accessible for percutaneous injection. Patients who are scheduled for surgical biopsy or tumor resection surgery will be injected 4 to 72 hours prior to surgery using the CIVO device. Minute volumes (up to 8.3 microliters) of saline (negative control) or microdoses of anti-cancer agents will be percutaneously injected in a columnar fashion through each of 8 needles into a single solid tumor. Following the patient's biopsy surgery or tumor resection surgery, the injected portion and a small uninjected portion will be used to determine the in situ drug response in the tumor. None of the data from this evaluation will be shared with patients or used to make clinical decisions. Study clinicians will have access to the patient's health record for 1 year after the study to monitor patient treatment responses. Such information will be used to help evaluate the correlation between clinical response and tumor response assessed via CIVO.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or over.
* At least one suspected soft tissue sarcoma tumor that is considered by the investigator to be: (1) accessible for percutaneous injection and (2) at least 2.5 cm in shortest dimension for patients undergoing an incisional biopsy, or at least 3 cm in shortest dimension for patients undergoing an excisional biopsy/tumor resection. Tumors should not be selected if the Investigator believes them to be necrotic or exhibit signs of radiation-induced fibrosis.
* Prior surgical evaluation and plan for surgical biopsy or surgery to remove the tumor being injected.
* ECOG performance status of 0-2 (or a Karnofsky performance status of >50%)
* Labs required for enrollment (prior to microinjection):

  * Absolute neutrophil count > 1000/mm3
  * Platelet count > 50,000/mm3
  * Hematocrit > 25%
  * Creatinine <3.0 mg/dl
  * Total Bilirubin <4.0 mg/dl
  * Bilirubin <4.0 mg/dl, SGOT ≤ 1.5 times the upper limit of normal
  * PT and PTT ≤ 1.5 times the upper limit of normal

Exclusion Criteria:

* Subjects with active fungal, viral, or bacterial infections.
* Pregnant women.
* Inability to give informed consent.
* Current treatment with anticoagulation such as warfarin or low-molecular-weight heparin.
* Tumors near critical structures such as those located near or in the brain or spine. This assessment will be determined by the treating clinician.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2016-12-15 (Actual); Primary Completion 2021-07-22 (Actual); Study Completion 2021-09-22 (Actual)

PRIMARY OUTCOMES:
Quantification of fraction of cells positive for apoptosis and drug target engagement biomarkers around injected drugs | 4-72 hours after microinjection
  Analysis will be performed to determine if there is a difference in responses caused by each drug versus the vehicle control

SECONDARY OUTCOMES:
Number of patients with adverse events related to pain | up to 28 days after microinjection
  Relationship of AE to study device or study procedure will be determined using an AE Relatedness Grading System.
Coefficient of variation and intra-class correlation coefficient of fraction of cells around injected drug in multiple tumor planes | 4-72 hours after microinjection
  Analysis will be performed for fraction of cells positive for apoptosis and drug target engagement biomarkers

CONTACTS AND LOCATIONS:
Overall Officials: Gary Deutsch, MD, Principal Investigator — Northwell Health; Kenneth Gundle, MD, Principal Investigator — Oregon Health & Science University (OHSU); Seth Pollack, MD, Principal Investigator — Fred Hutchinson Cancer Research Center/SCCA
Locations (3):
- United States (3):
  - Monter Cancer Center (Northwell Health), Lake Success, New York
  - OHSU Knight Cancer Institute, Portland, Oregon
  - Fred Hutchinson Cancer Research Center/Seattle Cancer Care Alliance (SCCA)/University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gundle KR, Deutsch GB, Goodman HJ, Pollack SM, Thompson MJ, Davis JL, Lee MY, Ramirez DC, Kerwin W, Bertout JA, Grenley MO, Sottero KHW, Beirne E, Frazier J, Dey J, Ellison M, Klinghoffer RA, Maki RG. Multiplexed Evaluation of Microdosed Antineoplastic Agents In Situ in the Tumor Microenvironment of Patients with Soft Tissue Sarcoma. Clin Cancer Res. 2020 Aug 1;26(15):3958-3968. doi: 10.1158/1078-0432.CCR-20-0614. Epub 2020 Apr 16. PMID 32299817